CLINICAL TRIAL: NCT05626686
Title: An Exploratory Investigation of the Effects of Single Use vs. Reuse Catheters in Intermittent Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CP352
Record Dates: First submitted 2022-08-25; First posted 2022-11-25 (Actual); Results first posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2023-10

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: The investigation is designed as an open-labelled, single-arm investigation including subjects currently using single use catheters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CLINY reusable catheter 28 days (Experimental): The investigation is designed as an open-labelled, single-arm investigation, in which the reuse CLINY catheter will be compared to single use catheters at baseline.
  Interventions: Device: CLINY catheter

INTERVENTIONS:
Device: CLINY catheter — Subjects using a single use catheter for bladder management at inclusion. During the study period, subjects will use the reusable CLINY catheter for 28 test-days

SUMMARY:
The overall aim of the investigation is to investigate the effect of repeated reuse of intermittent urinary catheters and to observe the impact of switch from single use to multiple reuse catheters.

DETAILED DESCRIPTION:
Throughout the investigation, the impact of switch from single use to multiple reuse catheters will be observed and compared with respect to health-related quality of life (HR-QoL), satisfaction, perception, and preference in female and male catheter-users, who use clean intermittent catheterization (CIC) for bladder management.

Furthermore, the investigation intends to identify microbial contamination of reused catheters and compare proportions to a control single use catheter.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age and has full legal capacity
2. Signed informed consent form
3. Use clean intermittent catheterization to the greatest extent possible (at least three times daily) for at least the last 1 month prior to inclusion
4. Ability (assessed by the investigator) and willingness to participate in a 4-week study period with at least three catheterizations a day using the investigational test product
5. Self-catheterize using a single use hydrophilic coated catheter for at least 1 month prior to inclusion

Exclusion Criteria:

1. Participation in any other clinical intervention study during this investigation
2. Previous participation in this investigation
3. Any known allergies towards ingredients in the investigational device
4. Symptoms of UTI at time of inclusion, as judged by the investigator
5. Antibiotic treatment within 2 weeks prior to the Baseline visit (V1)
6. Pregnancy
7. Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Andersen, Principal Investigator — Odense Universitetshospital; Nessn Azawi, Principal Investigator — Zealand University Hospital; Brian Kloster, Principal Investigator — Ålborg Universitetshospital
Locations (1):
- Odense Universitetshospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CLINY Reusable Catheter: Subjects used the reusable CLINY catheter for 28 days, replacing their regular use of single-use catheters.
Period: Overall Study
Arm/Group | CLINY Reusable Catheter
Started | 39
Completed | 33
Not Completed | 6
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | CLINY Reusable Catheter
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 33
Height, Continuous [Mean (Standard Deviation); unit: Centimeters] | 175.3 (10.0)
Weight, Continuous [Mean (Standard Deviation); unit: Kilograms] | 81.5 (17.3)
Reason for IC use, Categorical [Count of Participants; unit: Participants]
  Spinal Cord Injury | 4
  Multiple Sclerosis | 8
  Benign Prostatic Hyperplasia | 4
  Poor bladder emptying | 11
  Other | 6
Right hand function, Categorical [Count of Participants; unit: Participants]
  Normal dexterity | 29
  Reduced dexterity | 4
Left hand function, Categorical [Count of Participants; unit: Participants]
  Normal dexterity | 25
  Reduced dexterity | 6
  Do not know | 2
Urethral Sensitivity, Categorical [Count of Participants; unit: Participants]
  Impaired | 4
  Normal | 24
  None | 5
Time since starting IC as bladder management method, Continuous (years) [Mean (Standard Deviation); unit: years] | 9.2 (10.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Health-related Quality of Life From Baseline (Visit 1) to Termination (Visit 5), Measured by the Intermittent Self-Catheterization Questionnaire Index Score.
Description: The Intermittent Self-Catheterization Questionnaire is a validated, self-reported questionnaire which is scored on a 5-point Likert scale and is translated to a value ranging from 0 (strongly disagree) to 4 (strongly agree) with higher values corresponding to greater Health-related Quality of Life. The aggregate scores across domains and the total score are calculated by averaging and multiplying by 25 to achieve a 100-point scale. Change = (Termination score - Baseline score)
Time Frame: Baseline (day 0) and Termination (day 28).
Population: The full analysis set constituted all subjects enrolled who had been exposed to at least one device, with at least one endpoint recorded (data non-missing).
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CLINY Reusable Catheter
Number analyzed (Participants) | 33
score on a scale
  Baseline visit | 79.09 [73.69 to 84.49]
  Termination visit | 56.66 [51.26 to 62.06]

2. Secondary Outcome: Adverse Events
Description: Number of Adverse Events during the study
Time Frame: 28 days
Population: as for outcome 1
Measure: Number; unit: Adverse events
Arm/Group | CLINY Reusable Catheter
Number analyzed (Participants) | 33
Adverse events | 11

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | CLINY Reusable Catheter
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 8/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CLINY Reusable Catheter (N=39)
Blood in urine (Renal and urinary disorders) | 5 (5)
Urinary Tract Infection (Renal and urinary disorders) | 4 (4)
Tears in the urethra (Renal and urinary disorders) | 1 (1)
Pain in urinary tract (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/86/NCT05626686/Prot_SAP_000.pdf